CLINICAL TRIAL: NCT05460598
Title: The Effect of Cooling With a Bed Topper and Linen on Itch in Clinical Routine - an Exploratory Study
Brief Title: The Effect of Cooling With a Bed Topper and Linen on Itch in Clinical Routine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-00160; th21Mueller2
Record Dates: First submitted 2022-07-04; First posted 2022-07-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Itch
Keywords: cooling beddings; sleep quality; scratching; itch reduction; itch; nocturnal
MeSH Terms: conditions — Pruritus; Sleep Initiation and Maintenance Disorders | interventions — Bedding and Linens

STUDY DESIGN:
Intervention Model Description: Single-center, investigator-initiated, single-blinded, interventional, exploratory study.
Who Masked: Participant
Masking Description: single-blinded (only patients blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group: beddings with cooling effects (Active Comparator): Cooling beddings: linen made of the Outlast Technology https://www.outlast.com/en/. This product is made of 100 % lyocell and utilizes phase change materials based on natural wax. When this phase change material melts, heat is extracted from the environment and stored in microcapsules called thermocules. When the body cools down, these thermocules harden again release the heat from the linen. This might help to balances the body temperature and prevent warmth-aggravated itch.
  - The mattress is made of polyurethane foam and designed as a "cool gel" topper to be placed onto the standard hospital mattress. Heat is also absorbed and stored into this topper. This topper is covered with an Obatex cover. It protects the "cool gel" topper from moisture and organic liquids and is made of polyamide fabric.
  Interventions: Other: beddings with cooling effects
- control group: commonly used bedding (Placebo Comparator)
  Interventions: Other: commonly used bedding

INTERVENTIONS:
Other: beddings with cooling effects — beddings with cooling effects (mattress topper and bed linen)
  Arms: interventional group: beddings with cooling effects
Other: commonly used bedding — commonly used bedding
  Arms: control group: commonly used bedding

SUMMARY:
This single-blinded (only patients blinded) study is to assess the effect of cooling beddings on itch.

The primary objective is to test whether or not the use of the cooling beddings during 3 days can add at least 20% improvement in (nocturnal) itch as measured by the 0-10 NRS in comparison to a control group that does not use the cooling beddings.

DETAILED DESCRIPTION:
Itch is the most common skin-related symptom. Staying/sleeping in a bed with a cooling properties could have a positive effect on (nocturnal) itch intensity, sleep quality and daytime performance in consequence. A mattress topper and bed linen with cooling effects that are commercially available (https://www.oba.ch/cool_gel_topper) by the OBA AG (Basel), which is the supplier of beds and bedding items of the University Hospital Basel, has been used in clinical routine. This single-blinded (only patients blinded) study is to assess the effect of cooling beddings on itch and to better rationalize the beddings 'use. No comparative data is available and the design is purely exploratory. The primary objective of this study is to test whether or not the use of the cooling beddings during 3 days can add at least 20% improvement in (nocturnal) itch as measured by the 0-10 NRS in comparison to a control group that does not use the cooling beddings.

ELIGIBILITY:
Inclusion Criteria:

* Mean itch intensity NRS > 5 in the past 3 days
* Literacy and ability to read
* Inpatient stay required for > 3 nights

Exclusion Criteria:

* Age < 18 years
* Illiteracy
* Cognitive impairment (exclusion in case of mild cognitive impairment according to the Montreal-Cognitive Assessment (MOCA))
* The duration of the hospitalisation is foreseen to be shorter than 3 days
* Para- and Tetraplegia
* Hemisensory syndrome
* Core body temperature >38°C
* Use of other bedding > 8 hours or 2nd time request
* Use of an occlusive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
improvement in (nocturnal) itch | NRS ratings will be assessed every 6 hours (throughout 72 hours)
  improvement in (nocturnal) itch as measured by the 0-10 Numeric rating Scale (NRS) (at least 2 NRS points per 24 hours to obtain a meaningful therapeutic benefit). (NRS, 0= no itch, 10= worst imaginable)

SECONDARY OUTCOMES:
Scratching activity measured by actigraph (Actigraph qGT3X-BT) on the dominant wrist | Continuously recorded throughout 72 hours
  Comparison of the actigraphy of the interventional versus control group.to record hand movements as a surrogate marker for scratching activity and to record sleep tracking functions.
Richards-Campbell-Sleep Questionnaire (RCSQ) after each of the three nights addressing the sleep quality | Assessment after each night (3 times, altogether 72 hours)
  Sleep quality assessment by RCSQ. It consists of six items addressing "Sleep depth", "Sleep latency", "Awakenings", "Returning to sleep", "Sleep quality" and "Noise", each of which is rated on a visual analogue scales ranging from 0-100 mm. A higher value of the average score represents better sleep.
Patient questionnaire (regarding lying comfort, cooling pleasantness) | One time assessment after the third night
  Patient questionnaire regarding lying comfort, cooling pleasantness (5-point Likert scales, items "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree" and "Strongly agree")
Patient questionnaire regarding cooling intensity | One time assessment after the third night
  Patient questionnaire regarding cooling intensity (0-10/ no cooling- strongest-possible cooling).
Staff questionnaire regarding time practicability | Assessment after staff shift (3 times, altogether 72 hours)
  Staff questionnaire regarding time practicability (putting on/of the linen, weight of topper, cleaning procedure of cooling beddings) (5-point Likert scales: "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree" and "Strongly agree") after their shift.
Vital signs measured by Fitbit tracker | Continuously recorded throughout 72 hours
  On the non-dominant wrist, patients will wear a tracker (Fitbit Charge 5, Fitbit LLC, USA) to capture vital signs (e.g. heart rate, respiratory rate and skin temperature).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mueller, PD Dr. med., Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland